CLINICAL TRIAL: NCT05500937
Title: Effect of UDCA on the New Onset Diabetes and Glucose Intolerance Induced by Statin-A Multicenter, Prospective, Random Controlled Trial
Brief Title: Effect of UDCA on the New Onset Diabetes and Glucose Intolerance Induced by Statin
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XJTU1AF2021CRF-007
Record Dates: First submitted 2021-12-10; First posted 2022-08-15 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UDCA 500mg per day (Active Comparator): This group of participants receive UDCA 500mg per day.
  Interventions: Drug: UDCA
- Placebo (Placebo Comparator): This group of participants receive placebo.
  Interventions: Drug: UDCA

INTERVENTIONS:
Drug: UDCA — UDCA vs. placebo together with statin in ASCVD patients
  Other Names: Ursodeoxycholic acid

SUMMARY:
At present, it is recognized that statins are the cornerstone of treatment for the prevention of major cardiovascular events in patients with atherosclerotic cardiovascular disease (ASCVD); However, at the same time, the increased risk of long-term glucose tolerance and type 2 diabetes mellitus caused by statin therapy has attracted wide attention. The investigators' recent study found that the levels of glycosylated hemoglobin, insulin and C-peptide increased significantly with the extension of follow-up time in patients with hyperlipidemia. At the same time, serum and fecal bile acid metabolism profiles, especially secondary bile acid metabolism, were extensively changed, especially in ursodeoxycholic acid (UDCA), suggesting that the decrease of UDCA is a possible mechanism for statins to induce side effects of diabetes. According to this hypothesis, ursodeoxycholic acid combined with statins may improve the abnormal glucose tolerance caused by statins and maximize the benefit of statins. This study is a multicenter, prospective, randomized, parallel, double-blind placebo-controlled, cohort study. Taking ASCVD patients as the research object, the investigators will compare the changes of glycosylated hemoglobin, fasting blood glucose, fasting insulin, C-peptide and metabolomic indexes before and after the use of ursodeoxycholic acid combined with atorvastatin and atorvastatin alone and during follow-up, Further evaluate the changes of blood glucose related indexes before and after the use of ursodeoxycholic acid combined with atorvastatin and atorvastatin alone, clarify the possible mechanism and specific treatment targets of abnormal glucose tolerance caused by statin, and put forward a possible alternative treatment for the disorder of glucose metabolism caused by statin.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old and < 80 years old, regardless of gender;
* For those who had indications for taking statins for more than half a year, glycosylated hemoglobin increased by more than 0.5 and > 6.1% compared with half a year ago;
* Agree to accept the study treatment plan and voluntarily sign the informed consent form.

Exclusion Criteria:

* previous diagnosis of diabetes mellitus;
* Received hypoglycemic drug treatment;
* The level of abdominal blood glucose at baseline was ≥ 7mmol / L;
* Need to take glucocorticoids for a long time;
* Acute myocardial infarction and stroke occurred in the last 6 months;
* Severe liver dysfunction;
* Glomerular filtration rate (EGFR) < 30ml / min / 1.73m2 (MDRD formula);
* Malignant tumor;
* Blood system diseases;
* Acute or severe systemic infection;
* Women during pregnancy, lactation and preparation for pregnancy;
* Alcohol and other drug addicts and mental patients;
* Patients who are participating in other clinical studies or withdraw from less than 1 month;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of HbA1c | 12 months after enrollment
  Changes of glycosylated hemoglobin after taking ursodeoxycholic acid for half a year

SECONDARY OUTCOMES:
Concentration of blood lipid | 12 months after enrollment
Concentration of fasting blood glucose | 12 months after enrollment
Concentration of fasting islets | 12 months after enrollment
Concentration of bile acids | 12 months after enrollment
Rate of MACE | 12 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Zuyi Yuan, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided